CLINICAL TRIAL: NCT07188207
Title: The Efficacy of Adding Preoperative Rectal Misoprostol for Decreasing Intraoperative and Postoperative Blood Loss at Elective Cesarean Section
Brief Title: Rectal Misoprostol for Reducing Blood Loss in Elective Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Zanaty Khalaf Abbas, Resident, Obstetric and Gynecology Department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MISOCS-2025
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Misoprostol; Oxytocin; Cesarean Delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two equal parallel groups: one receiving oxytocin alone (control group), and the other receiving oxytocin plus rectal misoprostol (intervention group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be conducted in a blinded manner. Neither the participants nor the outcome assessors will know the treatment allocation. Care providers administering the intervention will also be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Oxytocin only (Experimental): Description: Participants receive standard intraoperative uterotonic therapy with oxytocin according to hospital protocol immediately after delivery of the baby and placenta. Standard perioperative care (spinal anesthesia, prophylactic antibiotics, fluid management, monitoring) is provided. Rescue uterotonic measures and transfusion given as clinically indicated.
  Interventions: Drug: Oxytocin
- Intervention: Oxytocin + Rectal Misoprostol (Experimental): Participants receive the same oxytocin regimen as Arm 1 plus a single rectal dose of misoprostol (600-1000 µg depending on risk profile) administered immediately after delivery of the baby and placenta. Standard perioperative care is identical to Arm 1. Rescue uterotonic measures and transfusion given as clinically indicated.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intravenous oxytocin administered per hospital protocol immediately after delivery of the baby and placenta (example regimen: 10 IU slow IV bolus followed by infusion e.g., 20 IU in 500-1000 mL isotonic crystalloid run over 2-4 hours; actual dosing adjusted per anesthesiologist/obstetrician and hospital policy). Document exact time, dose, and infusion rate in each case.
  Single rectal dose of misoprostol 600-1000 µg (select dose based on patient risk profile; e.g., 600 µg for routine prophylaxis, 800-1000 µg for high-risk cases) inserted into the rectum immediately after delivery of the baby and placenta. No dilution required.

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of adding preoperative rectal misoprostol to standard oxytocin for reducing intraoperative and postoperative blood loss in women undergoing elective cesarean section. Misoprostol is a prostaglandin E1 analogue that is inexpensive, heat-stable, and effective as a uterotonic agent. The study will compare outcomes between two groups: women receiving oxytocin alone and women receiving oxytocin plus rectal misoprostol. The primary outcome is the reduction of blood loss during and after surgery. Secondary outcomes include changes in hemoglobin levels, need for additional uterotonics, maternal safety, and overall recovery.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a leading cause of maternal morbidity and mortality worldwide, with increased risk following cesarean section compared to vaginal delivery. Oxytocin is the standard uterotonic agent used to prevent PPH, but it has several limitations including the need for refrigeration and potential cardiovascular side effects when administered rapidly.

Misoprostol, a prostaglandin E1 analogue, has gained attention as an effective alternative or adjunct to oxytocin because it is heat-stable, inexpensive, widely available in tablet form, and can be administered by various routes. The rectal route is particularly advantageous, providing rapid absorption, sustained uterine contraction, and fewer gastrointestinal side effects. However, its onset of action is slower than oxytocin, which may affect intraoperative hemostasis if uterine tone is not achieved quickly.

This study is designed as a randomized controlled trial conducted at the Department of Obstetrics and Gynecology, Assiut University Hospital. Eligible participants will be women aged 18-45 years with singleton pregnancies at ≥37 weeks of gestation undergoing elective cesarean section. Participants will be randomized into two groups:

Group A (Control): Oxytocin only, given according to hospital protocol immediately after delivery of the baby and placenta.

Group B (Intervention): Oxytocin plus a single rectal dose of misoprostol (600-1000 µg, based on risk profile) administered immediately after delivery of the baby and placenta.

The primary outcome will be the reduction in intraoperative and postoperative blood loss. Secondary outcomes will include changes in pre- and postoperative hemoglobin levels, need for additional uterotonic agents, maternal safety, ease and feasibility of rectal administration, and postoperative recovery.

The total sample size is 282 participants (141 per group), calculated to provide 80% power at a 95% confidence level to detect a significant reduction in blood loss. Data will be analyzed using SPSS software, with chi-square and independent sample t-tests applied as appropriate. Statistical significance will be considered at p < 0.05.

This trial seeks to provide evidence on the effectiveness and practicality of rectal misoprostol as an adjunct to oxytocin for reducing maternal blood loss during elective cesarean section, potentially improving outcomes and cost-effectiveness, particularly in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years.
* Singleton pregnancy at ≥37 weeks of gestation.
* Elective cesarean section planned under spinal anesthesia.
* Hemodynamically stable prior to surgery.
* Provided written informed consent.

Exclusion Criteria:

* Multiple pregnancy.
* Antepartum hemorrhage (e.g., placenta previa, abruption).
* Coagulopathy, thrombocytopenia, or anticoagulant therapy.
* Severe medical comorbidities (e.g., uncontrolled hypertension, cardiac disease, hepatic or renal impairment).
* Known allergy or contraindication to prostaglandins or oxytocin.
* Intrauterine fetal death or major fetal anomaly.
* Refusal to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 282 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative and postoperative blood loss | From skin incision until 24 hours after cesarean delivery
  Total blood loss will be measured intraoperatively by suction canister volume (minus irrigation fluid) and gravimetric method (weighing surgical pads/swabs), and postoperatively by weighing perineal pads up to 24 hours.

SECONDARY OUTCOMES:
Change in Hemoglobin and Hematocrit | Preoperative (within 24 hours before surgery) and 24 hours postoperative
  Difference between pre- and postoperative hemoglobin/hematocrit values to estimate blood loss.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Federspiel JJ, Eke AC, Eppes CS. Postpartum hemorrhage protocols and benchmarks: improving care through standardization. Am J Obstet Gynecol MFM. 2023 Feb;5(2S):100740. doi: 10.1016/j.ajogmf.2022.100740. Epub 2022 Sep 2. PMID 36058518